CLINICAL TRIAL: NCT04922788
Title: a Phase 3, Adaptive, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Immunogenicity, and Efficacy of the Nanocovax Vaccine Against COVID-19 in Volunteer Subjects 18 Years of Age and Older.
Brief Title: Study to Evaluate the Safety, Immunogenicity, and Efficacy of Nanocovax Vaccine Against COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NNG27
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 mcg Dose (Experimental): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Nanocovax
- Placebo (Placebo Comparator): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nanocovax — Recombinant Protein spike (s) SARS-CoV-2 and 0,5 mg Aluminum adjuvant
  Arms: 25 mcg Dose
Biological: Placebo — 0,5 mg Aluminum adjuvant
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity, and efficacy of Nanocovax vaccine in volunteer subjects 18 years of age and older.

DETAILED DESCRIPTION:
This is a phase 3, adaptive, multicenter, randomized, double-blind, placebo control study to evaluate the safety, immunogenicity, and efficacy of the Nanocovax vaccine against COVID-19 in volunteer subjects 18 years of age and older.

Age stratified as 18-45, 45-60, and > 60 years of age.

The assessment of immunogenicity will be further expanded in a subset of Phase 3 (1000 participants).

Randomly assigned to vaccine or placebo group with a ratio of 2:1 (2 subjects injected with Nanocovax 25 mcg : 1 subject injected with placebo).

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female 18 years of age or older.
* For females: Be of non-childbearing potential or willing to use appropriate contraceptive measures for 30 days prior to vaccination through 6 months after completion of the vaccine series.
* Willingness to provide a signed, printed, and dated informed consent form.
* Able and willing to participate in all activities in the clinical trial.
* Participants with HIV, HBV, HCV should have a health record, determined to be stable for 6 months prior to the screening.

Exclusion Criteria:

* Participants with unstable pre-existing medical conditions over the three months before enrollment (condition that has worsened to require hospitalization or significant changes in therapy).
* Planned administration/administration of a vaccine not foreseen by the study protocol from within 45 days before the first dose of study vaccine.
* Previous vaccination with any Covid-19 vaccine.
* History of COVID-19 disease.
* History of allergic reactions or anaphylaxis to previous immunizations or allergies to any components of the vaccine.
* Planning to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase through 6 months after the second immunization.
* History of bleeding disorders/hemostasis or use of anticoagulants.
* Currently having cancer or undergoing cancer treatment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 3 months prior to the first vaccine dose (inhaled and topical steroids are allowed).
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13006 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience a first episode of virologically-confirmed {reverse transcription polymerase chain reaction (RT-PCR) positive} case of COVID-19 of any severity | From 14 days after the second dose of study intervention to the end of the study, up to 1 year
  Per 1000 person-years of follow-up
Percentage of participants reporting Serious adverse events or medically attended adverse events | From dose 1 through one year after the last dose
Geometric mean of Anti-S IgG concentrations at each time point in a subset of participants | days 0, 42, 180, 365 after vaccination
Geometric mean of SARS-CoV-2 serum neutralizing titers by Plaque reduction neutralization test (PRNT) at each time point in a subset of participants | days 0, 42 after vaccination

SECONDARY OUTCOMES:
Percentage of participants reporting solicited local and systemic reactions | 7 days after each study vaccination
Percentage of participants reporting unsolicited vaccine-related ≥ Grade 2 adverse events | 28 days after each study vaccination
Proportion of participants achieving ≥4-fold rise of Anti-S IgG at each time point in a subset of participants | days 0,42, 180, 365 after vaccination
T-cell responses (intracellular cytokine staining) | days 0, 42 after vaccination
  Change from baseline in the cell-mediated immune response in a subset of participants
Number of participants who experience a first episode of virologically-confirmed {reverse transcription polymerase chain reaction (RT-PCR) positive} asymptomatic case of COVID-19 | From 14 days after the second dose of study intervention to the end of the study, up to 1 year
  Per 1000 person-years of follow-up
Number of participants who experience a first episode of virologically-confirmed {reverse transcription polymerase chain reaction (RT-PCR) positive} mild case of COVID-19 | From 14 days after the second dose of study intervention to the end of the study, up to 1 year
  Per 1000 person-years of follow-up
Number of participants who experience a first episode of virologically-confirmed {reverse transcription polymerase chain reaction (RT-PCR) positive} moderate to severe case of COVID-19 | From 14 days after the second dose of study intervention to the end of the study, up to 1 year
  Per 1000 person-years of follow-up
Number of participants who death due to covid-19 confirmed with (RT-PCR) positive | From 14 days after the second dose of study intervention to the end of the study, up to 1 year
  Per 1000 person-years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Nguyen, MD, Study Director — Medical Affairs Department
Locations (1):
- Military Medical Academy, Hanoi, Vietnam